CLINICAL TRIAL: NCT07078578
Title: Construction of a Machine Learning Prediction Model for Postoperative Delirium in Kidney Transplant Patients Based on Clinical Data
Brief Title: A Predictive Model for Postoperative Delirium in Kidney Transplant Patients
Status: Completed | Type: Observational
Sponsor: Hua Zheng (Other)
Responsible Party: Sponsor-Investigator, Hua Zheng, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: SXBQEMZK20250701
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation; Delirium - Postoperative; Cognitive
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium Group: Kidney transplant recipients who developed postoperative delirium within 7 days after surgery, identified through EMR text mining and structured data extraction.
- Non-Delirium Group: Kidney transplant recipients who did not develop postoperative delirium within 7 days after surgery.

SUMMARY:
This study aims to develop and prospectively validate a machine learning-based prediction model for postoperative delirium in kidney transplant recipients, using perioperative clinical data. Delirium is a common and serious postoperative complication that significantly increases morbidity, mortality, and healthcare costs. By analyzing electronic medical records from kidney transplant patients, including preoperative, intraoperative, and postoperative variables, the study seeks to identify high-risk patients and key predictors. Six machine learning models, including XGBoost, LGBM, GBC, LR, ANN, and SVM, will be constructed and evaluated, with a soft voting ensemble classifier used to optimize prediction performance. The goal is to improve early recognition and clinical management of postoperative delirium in kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent kidney transplantation at [Hospital Name, if needed] between January 1, 2016, and May 31, 2025.

Age ≥ 18 years at the time of transplantation.

Discharged alive from the hospital after surgery.

Complete perioperative clinical data available, including preoperative evaluations, intraoperative records, and postoperative documentation

Exclusion Criteria:

* Patients with documented pre-existing delirium or major neurocognitive disorder before surgery.

Simultaneous or multi-organ transplantation (e.g., kidney-pancreas).

Death within 7 days postoperatively.

Incomplete or missing key electronic medical records preventing outcome assessment.

Patients who withdrew consent for use of clinical data for research purposes (for prospective part).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult patients (aged 16 years and older) who underwent kidney transplantation at a single tertiary medical center between January 1, 2016, and May 31, 2025. The study includes retrospective data (2016-2024) for model development and prospective data (2025) for external validation. All included patients were discharged alive and had complete perioperative clinical data available for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium Within 7 Days After Kidney Transplantation | 7 days after surgery
  Postoperative delirium will be identified within 7 days of surgery through automated extraction and structured analysis of electronic medical record text fields, including progress notes, nursing records, and medication orders for sedatives or anxiolytics. Delirium will be categorized by onset time, severity, treatment, and recovery status.

IPD SHARING:
Plan to Share IPD: No
The dataset includes sensitive clinical information from kidney transplant patients. IPD will not be shared due to patient privacy concerns and institutional data use restrictions.